CLINICAL TRIAL: NCT01227967
Title: A Randomized Double-Blind Phase 2 Study Comparing the Efficacy, Safety, and Tolerability of Combination Antivirals (Amantadine, Ribavirin, Oseltamivir) Versus Oseltamivir for the Treatment of Influenza in Adults at Risk for Complications
Brief Title: Comparing the Efficacy, Safety, and Tolerability of Combination Antivirals (Amantadine, Ribavirin, Oseltamivir) Versus Oseltamivir for the Treatment of Influenza in Adults at Risk for Complications
Acronym: IRC003
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10-I-0210; 10-I-0210; IRC003
Record Dates: First submitted 2010-10-22; First posted 2010-10-25 (Estimated); Results first posted 2017-07-11 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Influenza
Keywords: Adaptive Design; At Risk; H1N1; Synergy; TCAD
MeSH Terms: conditions — Influenza, Human | interventions — Amantadine; Ribavirin; Oseltamivir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Combination Therapy (Experimental): Amantadine, Ribavirin, Oseltamivir
  Interventions: Drug: Amantadine, Ribavirin, Oseltamivir
- Oseltamivir monotherapy (Active Comparator): Oseltamivir
  Interventions: Drug: Oseltamivir

INTERVENTIONS:
Drug: Amantadine, Ribavirin, Oseltamivir — Subjects were prescribed the medication twice daily for 5 days, and each dose consisted of one capsule of Oseltamivir 75 mg, three capsules of Ribavirin 200 mg for total of 600 mg, and one capsule of Amantadine 100 mg.
  Arms: Combination Therapy
Drug: Oseltamivir — Subjects were prescribed the medication twice daily for 5 days, and each dose consisted of one capsule of Oseltamivir 75 mg.
  Arms: Oseltamivir monotherapy

SUMMARY:
Seasonal influenza is responsible for many hospitalizations and deaths each year, despite effective antiviral treatments. Some individuals have medical conditions such as heart or lung diseases that make them particularly at risk of severe influenza infections that may result in hospitalization or death. Oseltamivir (Tamiflu) is used most often to treat flu, but there are still many hospitalizations, complications, and deaths even with treatment. This study evaluated the use of combination antivirals (amantadine, oseltamivir, and ribavirin) compared to oseltamivir alone in the treatment of influenza in an at-risk population.

DETAILED DESCRIPTION:
Seasonal influenza is responsible for approximately 226,000 excess hospitalizations annually and despite effective antivirals causes significant morbidity and mortality (estimated 24,000-50,000 deaths each year in the United States alone). The influenza virus that emerged in 2009 (A/California/07/2009 H1N1) caused fewer deaths (12,000 flu-related deaths in the U.S) but in contrast to seasonal flu, nearly 90 percent of the deaths with the 2009 H1N1 occurred among people younger than 65 years of age. The CDC has defined an at-risk population that accounts for the majority of hospitalization and morbidity associated with influenza. This study evaluated the use of combination antivirals as compared to oseltamivir alone in the treatment of influenza in an at-risk population.

Subjects who met the CDC definition for being at-risk and that present with an influenza-like illness were screened for the study. Those subjects with a confirmatory test for influenza (rapid antigen or PCR) were randomized in a 1:1 manner to receive a blinded study treatment consisting of either the combination of amantadine, oseltamivir, and ribavirin or oseltamivir alone for 5 days. Clinical, virologic, and laboratory assessments on Days 1, 3, 7, 14, and 28 were used for both safety and efficacy analysis.

Design:

* Participants were screened with a physical examination and medical history, along with blood tests and throat swabs to confirm influenza infection.
* Eligible participants were randomly assigned to take either oseltamivir alone (the current standard treatment for influenza) or to take oseltamivir, amantadine, and ribavirin. Participants had additional blood samples and throat swabs taken at the start of the study, and were shown how to complete a study diary at home.
* Participants received a study medication kit containing the medication to take at home twice a day for 5 days.
* Participants returned, with the medication kit, to the clinic on days 1 (the first day after the start of the study), 3, 7, 14, and 28. The first visit took 2 to 3 hours, but each subsequent visit took approximately 1 to 2 hours. Additional blood samples and throat swabs were taken at these visits.

Pilot study:

Due to the lack of reliable data concerning the AUC virologic endpoint, an "external" pilot study was conducted in the first 47 patients randomized to identify a primary endpoint and method of analysis, and to possibly modify the sample size. To ensure no effect on the type I error rate, data from these 47 patients were excluded from the primary and secondary efficacy analyses but were used in other analyses of secondary objectives.

ELIGIBILITY:
* INCLUSION CRITERIA:

Enrollment (Screening)

1. Signed informed consent prior to initiation of any study procedures
2. Presence of an underlying medical condition(s) that might increase risk of complications from influenza
3. History of an influenza-like illness defined as:

   * One or more respiratory symptom (cough, sore throat, or nasal symptoms) AND
   * Either
   * Fever (subjective or documented >38 degrees C) OR
   * 1 or more constitutional symptom (headache, malaise, myalgia, sweats/chills or fatigue)
4. Onset of illness no more than 96 hours before screening defined as when the subject experienced at least one respiratory symptom, constitutional symptom, or fever
5. Willingness to have samples stored

Randomization

1. Signed informed consent
2. Presence of a medical condition(s) that had been associated with increased risk of complications from influenza

   * Age 65 years of age or older
   * Asthma
   * Neurological and neuro-developmental conditions (including disorders of the brain, spinal cord, peripheral nerve, and muscle such as cerebral palsy, epilepsy [seizure disorders], stroke, moderate to severe developmental delay, muscular dystrophy, or spinal cord injury) [though still able to provide informed consent per inclusion criteria #1]
   * Chronic lung disease (such as COPD and cystic fibrosis)
   * Heart disease (such as congenital heart disease, congestive heart failure, and coronary artery disease)
   * Blood disorders (excluding genetic causes of anemia, as noted in the exclusion criteria)
   * Endocrine disorders (such as diabetes mellitus)
   * Kidney disorders
   * Liver disorders
   * Metabolic disorders (such as inherited metabolic disorders and mitochondrial disorders)
   * Weakened immune system due to disease or medication (such as people with HIV/AIDS, or cancer, chronic steroids or other medications causing immune suppression)
   * BMI ≥ 40(kg/m²)
3. Onset of illness no more than 96 hours before screening defined as when the subject experienced at least one respiratory symptom, constitutional symptom, or fever
4. Positive test for influenza (either rapid antigen or PCR)

   - Results from influenza testing obtained for clinical indications within 12 hours before screening/enrollment may be used if available. Randomization may proceed in cases of discrepant results (one positive and one negative)
5. One of the following to avoid pregnancy:

   * Females who were able to become pregnant (i.e., are not postmenopausal, have not undergone surgical sterilization, and are sexually active with men) must agree to use at least 2 effective forms of contraception from the date of informed consent through 6 months after the last dose of study drug. At least one of the methods of contraception should be a barrier method
   * Males who had not undergone surgical sterilization and are sexually active with women must agree to use condoms plus have a partner use at least one additional effective form of contraception from the date of informed consent through 6 months after the last dose of study drug
6. Willingness to have samples stored

EXCLUSION CRITERIA:

(for Enrollment or Randomization)

1. Women who were pregnant or breast-feeding, and men whose female partner(s) was pregnant
2. Inability to take oral medication or a history of gastrointestinal malabsorption that would preclude the use of oral medication.
3. Hemoglobin < 10 g/dL
4. WBC < 1.5 times 10(9)/L
5. Neutrophils < 0.75 x 10(9)/L
6. Platelets < 50 x 10(9)/L
7. History of genetic hemoglobinopathy (e.g., thalassemia major or sickle cell anemia) or autoimmune hemolytic anemia
8. Received more than 2 doses of any antiviral influenza medications since onset of influenza symptoms
9. Received stavudine (d4T), didanosine (ddI), zidovudine (AZT), or azathioprine within 30 days prior to study entry
10. Creatinine clearance less than 60 mL/min (estimated by the Cockcroft-Gault equation using serum creatinine)
11. History of autoimmune hepatitis
12. Uncompensated liver disease (defined as AST > 3 times site upper limit of normal (ULN), ALT > 3 times ULN, or Direct Bilirubin > 2 times ULN)
13. Clinical signs of end-stage liver disease including jaundice, coagulopathy, portal hypertension, esophageal varices, ascites, peripheral edema, gastrointestinal bleeding, or encephalopathy
14. Chronic liver disease categorized as Child-Pugh class C (Child-Pugh score 10-15)
15. Known hypersensitivity to rimantadine, amantadine, ribavirin, oseltamivir, peramivir, or zanamivir
16. Received live attenuated virus vaccine (influenza or other) within 3 weeks prior to study entry
17. Use of any investigational drug within 30 days or 5 half-lives (whichever was longer) prior to study entry
18. Participation in other research protocols that would require more than 100 mL of blood to be drawn in any 4-week period that overlaps with this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 881 (Actual)
Dates: Start 2010-09; Primary Completion 2016-05-02 (Actual); Study Completion 2017-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Beigel, MD, Study Chair — Leidos Biomedical Research, Inc. in support of Clinical Research Section, LIR, NIAID, Natinal Institutes of Health; John Treanor, MD, Study Chair — University of Rochester
Locations (91):
- United States (69):
  - Simon Williamson Clinic, Birmingham, Alabama
  - East Valley Family Physicians, Chandler, Arizona
  - Thomas Lenzmeier Family Practice, Glendale, Arizona
  - Central Phoenix Medical Center, Phoenix, Arizona
  - WCCT Global LLC, Costa Mesa, California
  - Advanced Rx Clinical Research, Garden Grove, California
  - Torrance Clinical Research Institute, Inc., Lomita, California
  - University of Southern California, Los Angeles, California
  - University of California at San Diego, San Diego, California
  - Westlake Medical Research (CA), Thousand Oaks, California
  - Los Angeles BioMedical Research Institute, Torrance, California
  - Empire Clinical Research, Upland, California
  - University of Colorado, Aurora, Colorado
  - Centennial - IMMUNOe International Research, Centennial, Colorado
  - University of Florida, Gainesville, Florida
  - Best Quality Research Inc., Hialeah, Florida
  - San Marcus Research Clinic, Inc., Miami, Florida
  - Medical Consulting Center, Miami, Florida
  - Suncoast Research Group, LLC, Miami, Florida
  - University of Miami, Miami, Florida
  - DMI Research, Inc., Pinellas Park, Florida
  - Northwestern University, Chicago, Illinois
  - Sneeze, Wheeze & Itch Associates, LLC, Normal, Illinois
  - Ridge Family Practice, Council Bluffs, Iowa
  - University of Iowa, Iowa City, Iowa
  - Research Integrity, LLC, Owensboro, Kentucky
  - Horizon Research Group, of Opelousas, LLC, Eunice, Louisiana
  - Centex Studies Inc. - Dr. Seep, Lake Charles, Louisiana
  - NIH Clinical Center, Bethesda, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - UMass Medical School, Worcester, Massachusetts
  - Henry Ford Health Systems, Detroit, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Florissant Internists, Bridgeton, Missouri
  - Clinical Research Advantage/ Skyline Medical Center, Elkhorn, Nebraska
  - Prairie Fields Family Medicine, Fremont, Nebraska
  - Southwest Family Physicians, Omaha, Nebraska
  - New Jersey Medical School, Newark, New Jersey
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - James J. Peters, VA Medical Center, The Bronx, New York
  - University of North Carolina-Chapel Hill, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - Clinical Research Solutions - Dr. Panuto, Middleburg Heights, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Montgomery Medical, Smithfield, Pennsylvania
  - Health Concepts, Rapid City, South Dakota
  - Clinical Research Solutions - Dr. Bart, Columbia, Tennessee
  - Clinical Research Solutions - Dr. Slandzicki, Franklin, Tennessee
  - Clinical Research Solutions - Dr. Hoppers, Jackson, Tennessee
  - Holston Medical Group, Kingsport, Tennessee
  - Clinical Research Solutions - Dr. Rowe, Nashville, Tennessee
  - Clinical Research Solutions - Dr. Dar, Smyrna, Tennessee
  - University of Texas Tech Amarillo, Amarillo, Texas
  - Family Medicine Associates of Texas, Carrollton, Texas
  - 3rd Coast Research Associates, Corpus Christi, Texas
  - University of Texas at Houston, Houston, Texas
  - Centex Studies Inc. - Dr. Pouzar, Houston, Texas
  - Pioneer Research Solutions, Inc., Houston, Texas
  - Texas Tech HSC, Lubbock, Texas
  - Centex Studies Inc. - Dr. Garcia, Pharr, Texas
  - Village Health Partners, Plano, Texas
  - Endeavor Clinical Trials, San Antonio, Texas
  - Bandera Family Healthcare Research, San Antonio, Texas
  - University of Virginia, Charlottesville, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
- Argentina (8):
  - Instituto Medico Platense, La Plata, Buenos Aires
  - Hospital Houssay, Vicente López, Buenos Aires
  - Centro de Educación Médica e Investigaciónes Clínicas (CEMIC), Buenos Aires
  - Fundación del Centro de Estudios Infectológicos (FUNCEI), Buenos Aires
  - Hospital General de Agudos J. M. Ramos Mejía, Buenos Aires
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - Hospital Rawson, Córdoba
  - Instituto Centralizado de Asistencia e Investigación Clínica Integral (CAICI), Santa Fe
- Australia (7):
  - Holdsworth House Med Practice, Darlinghurst, New South Wales
  - Taylor Square Private Clinic, Darlinghurst, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Royal Brisbane, Herston, Queensland
  - Northside Clinic, Fitzroy North, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
- Mexico (3):
  - Instituto Nacional de Ciencias Médicas y Nutrición (INCMN) Salvador Zubirán, México
  - Hospital General y de Alta Especialidad "Dr. Manuel GEA Gonzalez", Tlalpan
  - Instituto Nacional de Enfermedades Respiratorias (INER), Tlalpan
- Thailand (4):
  - Siriraj Hospital, Mahidol University, Bangkoknoi, Bangkok
  - HIV-NAT, The Thai Red Cross AIDS, Patumwan, Bangkok
  - Srinagarind Hospital, Khon Kaen University, Muang, Changwat Khon Kaen
  - Bamrasnaradura Infectious Diseases Institute, Muang, Changwat Nonthaburi

REFERENCES:
- [Background] Thompson WW, Shay DK, Weintraub E, Brammer L, Cox N, Anderson LJ, Fukuda K. Mortality associated with influenza and respiratory syncytial virus in the United States. JAMA. 2003 Jan 8;289(2):179-86. doi: 10.1001/jama.289.2.179. PMID 12517228
- [Background] Monto AS. Vaccines and antiviral drugs in pandemic preparedness. Emerg Infect Dis. 2006 Jan;12(1):55-60. doi: 10.3201/eid1201.051068. PMID 16494718
- [Background] Moscona A. Oseltamivir resistance--disabling our influenza defenses. N Engl J Med. 2005 Dec 22;353(25):2633-6. doi: 10.1056/NEJMp058291. No abstract available. PMID 16371626
- [Derived] Beigel JH, Bao Y, Beeler J, Manosuthi W, Slandzicki A, Dar SM, Panuto J, Beasley RL, Perez-Patrigeon S, Suwanpimolkul G, Losso MH, McClure N, Bozzolo DR, Myers C, Holley HP Jr, Hoopes J, Lane HC, Hughes MD, Davey RT; IRC003 Study Team. Oseltamivir, amantadine, and ribavirin combination antiviral therapy versus oseltamivir monotherapy for the treatment of influenza: a multicentre, double-blind, randomised phase 2 trial. Lancet Infect Dis. 2017 Dec;17(12):1255-1265. doi: 10.1016/S1473-3099(17)30476-0. Epub 2017 Sep 22. PMID 28958678
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2010-I-0210.html
- See also: The DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Version 1.0, December 2004 (Clarification, August 2009). — https://rsc.tech-res.com/clinical-research-sites/safety-reporting/daids-grading-tables

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Outpatient or hospitalized participants at high risk for complications and morbidity, diagnosed with influenza by rapid antigen or PCR were recruited at 65 sites from 5 countries: 52 from the U.S., 2 from Australia, 3 from Mexico, and 4 each in Thailand and Argentina, between March 2011 to April 2016.
Pre-assignment Details: Eight hundred eighty-one subjects were enrolled per protocol (signed consent). Two hundred fifty-one subjects were excluded during screening and did not participate in any other aspect of the trial. Three subjects were randomized improperly because they were given study drug kit prior to the randomization.
Groups:
- Combination Therapy: Drug: Amantadine, Ribavirin, Oseltamivir
  Subjects were prescribed the medication twice daily for 5 days, and each dose consisted of one capsule of Oseltamivir 75 mg, three capsules of Ribavirin 200 mg for total of 600 mg, and one capsule of Amantadine 100 mg.
- Oseltamivir Monotherapy: Drug: Oseltamivir
  Subjects were prescribed the medication twice daily for 5 days, and each dose consisted of one capsule of Oseltamivir 75 mg.
Period: Overall Study
Arm/Group | Combination Therapy | Oseltamivir Monotherapy
Started | 314 | 316
Completed (Results were through database cutoff (10 November 2016) for efficacy analysis (through Day 28 visit)) | 298 | 303
Not Completed | 16 | 13
Not completed — Protocol Violation | 3 | 1
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 8 | 3
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Physician Decision | 0 | 1
Not completed — Never Started Treatment | 0 | 4
Not completed — Taking Additional Antiviral Drug | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent To Treat (ITT) Population: all participants who were randomized properly and who had received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Combination Therapy | Oseltamivir Monotherapy | Total
Number analyzed (Participants) | 314 | 312 | 626
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 4 | 5
  Between 18 and 65 years | 252 | 241 | 493
  >=65 years | 61 | 67 | 128
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 49.5 [37 to 61] | 49.5 [35.5 to 61] | 49.5 [36 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 187 | 198 | 385
  Male | 127 | 114 | 241
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 55 | 58 | 113
  Not Hispanic or Latino | 258 | 254 | 512
  Unknown or Not Reported | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 203 | 189 | 392
  Asian | 70 | 73 | 143
  Black or African American | 18 | 25 | 43
  American Indian | 1 | 2 | 3
  Race not available to clinic | 21 | 21 | 42
  Subject does not want to report | 1 | 1 | 2
  Subject does not know | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  Argentina | 12 | 10 | 22
  United States | 220 | 216 | 436
  Mexico | 17 | 18 | 35
  Australia | 0 | 2 | 2
  Thailand | 65 | 66 | 131
Influenza Diagnostic Test by Local Testing [Count of Participants; unit: Participants]
  RT-PCR/PCR | 33 | 30 | 63
  Rapid antigen test | 281 | 281 | 562
  Isothermal nucleic acid amplification technology | 0 | 1 | 1
Positive Influenza Test by Local Testing [Count of Participants; unit: Participants] | 314 | 312 | 626
Result of Influenza Test By Local Testing [Count of Participants; unit: Participants]
  Influenza A/H1N1 | 13 | 14 | 27
  Influenza A/H3N2 | 1 | 1 | 2
  Influenza A unsubtypable | 29 | 22 | 51
  Influenza A not typed | 180 | 180 | 360
  Influenza B | 75 | 80 | 155
  Influenza positive (unknown A or B) | 10 | 5 | 15
  Multiple types/subtypes | 6 | 10 | 16
Confirmed Influenza Infection Status By Central Testing [Count of Participants; unit: Participants]
  Yes | 230 | 224 | 454
  No | 84 | 88 | 172
Influenza Type/Subtype By Central Testing [Count of Participants; unit: Participants] — Influenza type/subtype by central lab testing was from site-collected swab on Day 0 (the first one if more than one was collected) and if that was missing, then from a Day -1 sample, if collected
  Participants
    Influenza A/H3N2 | 126 | 118 | 244
    Influenza A/H1N1 | 55 | 49 | 104
    Influenza B | 49 | 57 | 106
    Negative | 83 | 86 | 169
    Missing | 1 | 2 | 3
Quantitative PCR Viral Shedding [Median (Inter-Quartile Range); unit: log10 copies/mL] — Limit of detection (LOD)/lower limit of quantification (LLOQ) for Flu A and Flu B by qPCR is 3.2/3.9 and 3.4/4.0, respectively.
  Results <LOD were imputed as LOD; results >=LOD and <LLOQ were imputed as LLOQ, and results >ULOQ were imputed as ULOQ Population: The results are for the 454 participants with a confirmed positive test for influenza on a Day 0 sample from the central laboratory using a RT-PCR for influenza type and subtype.
  log10 copies/mL
    number analyzed (Participants) | 230 | 224 | 454
    (all) | 6.4 [5.6 to 7.2] | 6.7 [5.1 to 7.7] | 6.5 [5.4 to 7.4]
Presence of fever [Count of Participants; unit: Participants]
  Yes | 94 | 93 | 187
  No | 216 | 216 | 432
  Missing | 4 | 3 | 7
Symptom Score [Count of Participants; unit: Participants] — Symptoms were scored on a 4-point scale : 0=absent, 1=mild, 2=moderate, 3=severe
  Participants
    Cough: Absent | 18 | 14 | 32
    Cough: Mild | 68 | 86 | 154
    Cough: Moderate | 139 | 130 | 269
    Cough: Severe | 85 | 78 | 163
    Cough: Missing | 4 | 4 | 8
    Fatigue: Absent | 28 | 15 | 43
    Fatigue: Mild | 33 | 43 | 76
    Fatigue: Moderate | 117 | 105 | 222
    Fatigue: Severe | 132 | 145 | 277
    Fatigue: Missing | 4 | 4 | 8
    Feverishness: Absent | 70 | 62 | 132
    Feverishness: Mild | 61 | 68 | 129
    Feverishness: Moderate | 111 | 98 | 209
    Feverishness: Severe | 68 | 80 | 148
    Feverishness: Missing | 4 | 4 | 8
    Diarrhea: Absent | 231 | 253 | 484
    Diarrhea: Mild | 36 | 26 | 62
    Diarrhea: Moderate | 26 | 20 | 46
    Diarrhea: Severe | 15 | 10 | 25
    Diarrhea: Missing | 6 | 3 | 9
    Muscle aches: Absent | 44 | 30 | 74
    Muscle aches: Mild | 51 | 56 | 107
    Muscle aches: Moderate | 100 | 99 | 199
    Muscle aches: Severe | 115 | 124 | 239
    Muscle aches: Missing | 4 | 3 | 7
    Vomiting: Absent | 268 | 269 | 537
    Vomiting: Mild | 18 | 18 | 36
    Vomiting: Moderate | 16 | 12 | 28
    Vomiting: Severe | 6 | 9 | 15
    Vomiting: Missing | 6 | 4 | 10
    Headache: Absent | 60 | 55 | 115
    Headache: Mild | 76 | 81 | 157
    Headache: Moderate | 99 | 99 | 198
    Headache: Severe | 75 | 74 | 149
    Headache: Missing | 4 | 3 | 7
    Nausea: Absent | 197 | 198 | 395
    Nausea: Mild | 54 | 51 | 105
    Nausea: Moderate | 38 | 35 | 73
    Nausea: Severe | 19 | 24 | 43
    Nausea: Missing | 6 | 4 | 10
    Sore throat: Absent | 80 | 80 | 160
    Sore throat: Mild | 94 | 91 | 185
    Sore throat: Moderate | 102 | 91 | 193
    Sore throat: Severe | 34 | 47 | 81
    Sore throat: Missing | 4 | 3 | 7
    Stuffy nose: Absent | 82 | 66 | 148
    Stuffy nose: Mild | 62 | 68 | 130
    Stuffy nose: Moderate | 107 | 96 | 203
    Stuffy nose: Severe | 59 | 78 | 137
    Stuffy nose: Missing | 4 | 4 | 8
    Rhinorrhea: Absent | 77 | 54 | 131
    Rhinorrhea: Mild | 79 | 96 | 175
    Rhinorrhea: Moderate | 96 | 84 | 180
    Rhinorrhea: Severe | 56 | 74 | 130
    Rhinorrhea: Missing | 6 | 4 | 10
Overall Symptom Score [Median (Inter-Quartile Range); unit: units on a scale] — Overall symptom score was the sum of available scores for each of the 11 symptoms assessed (so ignoring missing values). The possible range of the overall symptom score is therefore 0 (no symptoms) to 44 (severe for all 10 symptoms). Participants with missing evaluations for all symptoms were given a missing overall symptom score.
  units on a scale | 15 [11 to 19] | 15 [11 to 19] | 15 [11 to 19]
Functional status [Count of Participants; unit: Participants]
  Vigorous activities: Limited a lot = 0 | 238 | 238 | 476
  Vigorous activities: Limited a little = 50 | 58 | 59 | 117
  Vigorous activities: Not limited at all = 100 | 14 | 12 | 26
  Vigorous activities: Missing | 4 | 3 | 7
  Moderate activities: Limited a lot = 0 | 167 | 171 | 338
  Moderate activities: Limited a little = 50 | 114 | 107 | 221
  Moderate activities: Not limited at all = 100 | 29 | 31 | 60
  Moderate activities: Missing | 4 | 3 | 7
  Lifting groceries: Limited a lot = 0 | 99 | 116 | 215
  Lifting groceries: Limited a little = 50 | 129 | 114 | 243
  Lifting groceries: Not limited at all = 100 | 82 | 79 | 161
  Lifting groceries: Missing | 4 | 3 | 7
  Climbing stairs: Limited a lot = 0 | 182 | 172 | 354
  Climbing stairs: Limited a little = 50 | 97 | 105 | 202
  Climbing stairs: Not limited at all = 100 | 31 | 32 | 63
  Climbing stairs: Missing | 4 | 3 | 7
  Climbing 1 flight: Limited a lot = 0 | 97 | 103 | 200
  Climbing 1 flight: Limited a little = 50 | 146 | 129 | 275
  Climbing 1 flight: Not limited at all = 100 | 67 | 77 | 144
  Climbing 1 flight: Missing | 4 | 3 | 7
  Bending or kneeling: Limited a lot = 0 | 89 | 82 | 171
  Bending or kneeling: Limited a little = 50 | 118 | 133 | 251
  Bending or kneeling: Not limited at all = 100 | 103 | 94 | 197
  Bending or kneeling: Missing | 4 | 3 | 7
  Walking > 1 mile: Limited a lot = 0 | 199 | 202 | 401
  Walking > 1 mile: Limited a little = 50 | 81 | 78 | 159
  Walking > 1 mile: Not limited at all = 100 | 30 | 29 | 59
  Walking > 1 mile: Missing | 4 | 3 | 7
  Walking blocks: Limited a lot = 0 | 169 | 177 | 346
  Walking blocks: Limited a little = 50 | 100 | 91 | 191
  Walking blocks: Not limited at all = 100 | 41 | 41 | 82
  Walking blocks: Missing | 4 | 3 | 7
  Walking a block: Limited a lot = 0 | 101 | 108 | 209
  Walking a block: Limited a little = 50 | 123 | 111 | 234
  Walking a block: Not limited at all = 100 | 86 | 90 | 176
  Walking a block: Missing | 4 | 3 | 7
  Bathing/dressing self: Limited a lot = 0 | 48 | 54 | 102
  Bathing/dressing self: Limited a little = 50 | 72 | 83 | 155
  Bathing/dressing self: Not limited at all = 100 | 190 | 172 | 362
  Bathing/dressing self: Missing | 4 | 3 | 7
Average Functional Status [Median (Inter-Quartile Range); unit: units on a scale] — Average functional status was calculated as the average of the ten items assessed (so ignoring missing values), scoring 0='yes, limited a lot', 50='yes, limited a little', 100='no, not limited at all'. The possible range of the functional status score is therefore 0 (worst possible status) to 100 (best possible status). Participants with missing evaluations for all items were given a missing average functional status.
  units on a scale | 35 [20 to 60] | 35 [15 to 55] | 35 [15 to 60]
Global assessment [Count of Participants; unit: Participants]
  Subject feels as good today as before flu: Yes | 9 | 7 | 16
  Subject feels as good today as before flu: No | 301 | 302 | 603
  Subject feels as good today as before flu: Missing | 4 | 3 | 7
  Subject functions as well today as before flu: Yes | 23 | 20 | 43
  Subject functions as well today as before flu: No | 287 | 289 | 576
  Subject functions as well today as before flu: Missing | 4 | 3 | 7
Complications of Influenza [Count of Participants; unit: Participants]
  Sinusitis: Yes | 11 | 14 | 25
  Sinusitis: No | 298 | 298 | 596
  Sinusitis: Unable to assess | 2 | 0 | 2
  Sinusitis: Missing | 3 | 0 | 3
  Otitis Media: Yes | 2 | 4 | 6
  Otitis Media: No | 307 | 308 | 615
  Otitis Media: Unable to assess | 2 | 0 | 2
  Otitis Media: Missing | 3 | 0 | 3
  Bronchitis/Bronchiolitis: Yes | 8 | 14 | 22
  Bronchitis/Bronchiolitis: No | 301 | 298 | 599
  Bronchitis/Bronchiolitis: Unable to assess | 2 | 0 | 2
  Bronchitis/Bronchiolitis: Missing | 3 | 0 | 3
  Pneumonia: Yes | 5 | 9 | 14
  Pneumonia: No | 304 | 303 | 607
  Pneumonia: Unable to assess | 2 | 0 | 2
  Pneumonia: Missing | 3 | 0 | 3
  Using antibiotic for other reasons: Yes | 20 | 21 | 41
  Using antibiotic for other reasons: No | 291 | 291 | 582
  Using antibiotic for other reasons: Unable to assess | 0 | 0 | 0
  Using antibiotic for other reasons: Missing | 3 | 0 | 3
Medical Conditions [Count of Participants; unit: Participants] — Medication conditions that may increase risk of complications from influenza which are used to determine eligibility for the study.
  Participants
    >= 65 years: Yes | 251 | 247 | 498
    >= 65 years: No | 63 | 65 | 128
    Asthma: Yes | 214 | 213 | 427
    Asthma: No | 100 | 99 | 199
    Neurological condition: Yes | 297 | 293 | 590
    Neurological condition: No | 17 | 19 | 36
    Chronic Lung disease: Yes | 297 | 291 | 588
    Chronic Lung disease: No | 17 | 21 | 38
    Heart disease: Yes | 284 | 273 | 557
    Heart disease: No | 30 | 39 | 69
    Blood disorder: Yes | 306 | 307 | 613
    Blood disorder: No | 8 | 5 | 13
    Endocrine: Yes | 227 | 224 | 451
    Endocrine: No | 87 | 88 | 175
    Kidney: Yes | 306 | 306 | 612
    Kidney: No | 8 | 6 | 14
    Liver disorder: Yes | 311 | 305 | 616
    Liver disorder: No | 3 | 7 | 10
    Metabolic: Yes | 302 | 304 | 606
    Metabolic: No | 12 | 8 | 20
    Weakened immune system: Yes | 270 | 266 | 536
    Weakened immune system: No | 44 | 46 | 90
    BMI >= 40: Yes | 240 | 261 | 501
    BMI >= 40: No | 74 | 51 | 125

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Virus Detectable by Quantitative PCR (qPCR) in Nasopharyngeal (NP) Swabs
Description: The central laboratory performed a qualitative PCR test on the NP sample from Day 0 in order to confirm influenza infection and to determine the influenza type and subtype. For participants with a positive influenza test result at Day 0 from this qualitative PCR testing, the laboratory then performed qPCR testing of subsequent samples to quantify viral shedding.
Time Frame: At Day 3
Population: The population analyzed was restricted to the 407 participants who had a confirmed positive test for influenza by qPCR in the central laboratory testing and were not in the pilot study for IRC003. 13 participants (5 in the Combination Therapy and 8 in the Oseltamivir Monotherapy) had missing endpoint samples so were excluded from the analysis.
Measure: Number; unit: percentage of participants analyzed
Arm/Group | Combination Therapy | Oseltamivir Monotherapy
Number analyzed (Participants) | 200 | 194
percentage of participants analyzed | 40 | 50
Statistical Analysis 1: Comparison: Combination Therapy vs Oseltamivir Monotherapy; Assuming that pooled percentage of participants with virus detectable by PCR at Day 3 is 50%, assuming that the Combination Therapy was better than the Oseltamivir Monotherapy and that the detectable rate in the Combination Therapy was 42.5% compared to 57.5% in the Oseltamivir Monotherapy (a 15% reduction), and assuming 10% subjects with missing qPCR at Day 3, in a two-sided, two-sample 0.05-level t- test with 546 participants combined across both arms, there was 90% power; Test type: Superiority or Other; p = 0.046, Z-test, 2-sided — P-value was not adjusted for multiple interim analyses; Comparison of randomized arms was based on the normal approximation to the binomial distribution; Mean Difference (Final Values) = -10, 95% CI 2-sided [-19.8 to -0.2], Standard Error of Mean 5 — The difference in percents was calculated as the percent detectable in the Combination Therapy minus the percent detectable in the Oseltamivir Monotherapy

2. Secondary Outcome: Number of Participants by Virus Detection Status
Description: Number of participants who had undetectable values (less than the limit of detection [LOD]), who had values between the LOD and the lower limit of quantification (LLOQ), and who had values ≥LLOQ
Time Frame: At Day 0, 3 and 7.
Population: The population analyzed is the Primary Efficacy Population (PEP), which included all participants who were randomized properly, had received at least one dose of study drug, and had influenza virus isolated and typed in the qualitative PCR evaluation at Day 0 from central laboratory testing.
Measure: Count of Participants; unit: Participants
Arm/Group | Combination Therapy | Oseltamivir Monotherapy
Number analyzed (Participants) | 230 | 224
Participants
  Day 0: >=LLOQ | 221 | 200
  Day 0: >=LOD, <LLOQ | 4 | 9
  Day 0: <LOD | 5 | 15
  Day 0: Missing | 0 | 0
  Day 3: >=LLOQ | 65 | 87
  Day 3: >=LOD, <LLOQ | 22 | 25
  Day 3: <LOD | 134 | 104
  Day 3: Missing | 9 | 8
  Day 7: >=LLOQ | 19 | 24
  Day 7: >=LOD, <LLOQ | 4 | 7
  Day 7: <LOD | 193 | 184
  Day 7: Missing | 14 | 9

3. Secondary Outcome: qPCR Viral Shedding
Description: Median, 25% and 75% percentile of the value of viral shedding (Results <LOD were imputed as the LOD value, and Results >= LOD, <LLOQ were imputed as the LLOQ value.)
Time Frame: At Day 0, 3 and 7
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Log10 copies/mL
Arm/Group | Combination Therapy | Oseltamivir Monotherapy
Number analyzed (Participants) | 230 | 224
Log10 copies/mL
  Day 0 | 6.4 [5.6 to 7.2] | 6.7 [5.1 to 7.7]
  Day 3 | 3.4 [3.2 to 4.2] | 3.9 [3.2 to 4.95]
  Day 7 | 3.2 [3.2 to 3.4] | 3.2 [3.2 to 3.4]

4. Secondary Outcome: Number of Participants Shedding Virus
Description: Number of participants with undetectable viral load at both Day 3 and Day 7; detectable at Day 3 and undetectable at Day 7; detectable at Day 7 (irrespective of whether or not detectable at Day 3).
Time Frame: At day 3 and 7.
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Combination Therapy | Oseltamivir Monotherapy
Number analyzed (Participants) | 230 | 224
Participants
  Undetectable at both Day 3 and 7 | 126 | 95
  Detectable at Day 3 and undetectable at Day 7 | 67 | 88
  Detectable at Day 7 | 23 | 30
  Missing result at Day 3 and/or Day 7 | 14 | 11

5. Secondary Outcome: Time to Alleviation of Influenza Clinical Symptoms.
Description: The assessed symptoms were cough, nasal obstruction (stuffy nose), sore throat, fatigue, headache, muscle aches, feverishness, rhinorrhea, nausea, vomiting, diarrhea. Duration of clinical symptoms is defined as the time from Day 0 to the first of two successive measurements at which all clinical symptoms are grade 0 (absent) or 1 (mild). A measurement is considered to be the 8AM or 8PM assessment during Days 0 to 7 (so two measurements are obtained per day) and then the daily assessment thereafter. Time will then be calculated in half-days through to Day 7. If a subject's first two assessments on (baseline assessment and first subsequent diary card assessment) satisfy this criterion, then the duration will be set to zero. For participants who did not have two successive records meeting this criterion, follow-up was censored for analysis purposes at the time of the last but one diary card record with symptoms evaluated.
Time Frame: From treatment initiation to Day 28
Population: The population analyzed is the Intention To Treat (ITT) Population, which included all participants who were randomized properly and who had received at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Combination Therapy | Oseltamivir Monotherapy
Number analyzed (Participants) | 314 | 312
Days | 4.5 [4.0 to 5.0] | 4.0 [3.5 to 4.5]

6. Secondary Outcome: Time to Absence of Fever
Description: Fever was considered present based on the diary cards if a subject reported a maximal temperature ≥38.0°C (for the period since the diary card was previously completed) or reported having taken an antipyretic drug (also for the period since the diary card was previously completed). Otherwise, fever was considered not present during the period since the diary card was previously completed, except that the evaluation was considered missing if either the temperature or the antipyretic drug use entry was not completed on the diary card. The duration of fever was defined as the time from Day 0 to the first of two successive assessments (through to Day 7) or to the first assessment (Day 8 onwards) at which no fever was present according to this definition.For participants who did not have two successive records meeting this criterion, follow-up was censored for analysis purposes at the time of the last but one diary card record with fever evaluated.
Time Frame: From treatment initiation to Day 28
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Combination Therapy | Oseltamivir Monotherapy
Number analyzed (Participants) | 314 | 312
Days | 0.5 [NA to NA] — Not estimable | 0.5 [NA to NA] — Not estimable

7. Secondary Outcome: Time to Resolution of All Symptoms AND Fever
Description: The assessed symptoms were cough, nasal obstruction (stuffy nose), sore throat, fatigue, headache, muscle aches, feverishness, rhinorrhea, nausea, vomiting, diarrhea. Fever was considered present based on the diary cards if a subject reported a maximal temperature ≥38.0°C (for the period since the diary card was previously completed) or reported having taken an antipyretic drug (also for the period since the diary card was previously completed). Time to resolution of all clinical symptoms and fever is defined as the time from Day 0 to the first of two successive measurements at which all clinical symptoms are grade 0 (absent) or 1(mild) and no fever >=38.0 C or antipyretic drug is reported. For participants who did not have two successive records meeting this criterion, follow-up was censored for analysis purposes at the time of the last but one diary card record with symptoms and fever evaluated.
Time Frame: From treatment initiation to Day 28
Population: The population analyzed is the Intention To Treat (ITT) Population, which includes all participants who were randomized properly and who had received at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Combination Therapy | Oseltamivir Monotherapy
Number analyzed (Participants) | 314 | 312
Days | 4.5 [4.0 to 5.0] | 4.5 [4.0 to 5.0]

8. Secondary Outcome: Time to Feeling as Good as Before the Onset of the Influenza Illness
Description: Time to feeling as good as before influenza is defined as time to the first of two successive 'yes' responses to the question of 'feeling as good as you did before you had the flu'.For participants who did not have two successive records meeting this criterion, follow-up was censored for analysis purposes at the time of the last but one diary card record with question answered.
Time Frame: From treatment initiation to Day 28
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Combination Therapy | Oseltamivir Monotherapy
Number analyzed (Participants) | 314 | 312
Days | 7.5 [7.0 to 7.5] | 6.5 [6.0 to 7.0]

9. Secondary Outcome: Time to Return to Pre-influenza Function
Description: Time to return to pre-influenza function is defined as the time from Day 0 to the first of two successive 'Yes' answers to the global assessment question 'Are you functioning as well as you were before you had the flu'.For participants who did not have two successive records meeting this criterion, follow-up was censored for analysis purposes at the time of the last but one diary card record with question answered.
Time Frame: From treatment initiation to Day 28
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Combination Therapy | Oseltamivir Monotherapy
Number analyzed (Participants) | 314 | 312
Days | 7.0 [6.0 to 7.5] | 6.0 [5.0 to 6.5]

10. Secondary Outcome: Time to Return of Physical Function to Pre-illness Leve
Description: Time to return of physical function to pre-illness level was defined as the time from Day 0 to the first of two successive measurements at which the physical function score equals or is better than the pre-illness score (obtained by recall at enrollment).For subjects who did not have two successive records meeting this criterion, follow-up was censored for analysis purposes at the time of the last but one diary card record with physical function evaluated.
Time Frame: From treatment initiation to Day 28
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Combination Therapy | Oseltamivir Monotherapy
Number analyzed (Participants) | 314 | 312
Days | 7.0 [6.0 to 8.0] | 6.0 [6.0 to 7.0]

11. Secondary Outcome: Percentage of Participants With Clinical Failure at Day 5
Description: Clinical failure at Day 5 is defined as the need for continued (non-study) antiviral use after Day 5.
Time Frame: From treatment initiation to Day 28
Population: as for outcome 5
Measure: Number; unit: percentage of participants analyzed
Arm/Group | Combination Therapy | Oseltamivir Monotherapy
Number analyzed (Participants) | 314 | 312
percentage of participants analyzed | 7.0 | 7.7

12. Secondary Outcome: Percentage of Participants Who Develop Bronchitis, Pneumonia, or Other Complications of Influenza After Day 0.
Description: Participants were assessed for the signs/symptoms suggestive of one of the following complications: Sinusitis, Otitis Media ,Bronchitis / Bronchiolitis, Pneumonia and antibiotic use for reason other than above.
Time Frame: From treatment initiation to Day 28
Population: The population analyzed is the Intention To Treat (ITT) Population, which included all participants who were randomized properly and who had received at least one dose of study drug. The categories in the table are not mutually exclusive (because some participants had multiple complications) and the last row of the table summarizes all incidents.
Measure: Number; unit: percentage of participants analyzed
Arm/Group | Combination Therapy | Oseltamivir Monotherapy
Number analyzed (Participants) | 314 | 312
percentage of participants analyzed
  Sinustis | 4.5 | 4.5
  Otitis Media | 0.3 | 1.0
  Bronchitis Bronchiolitis | 5.7 | 3.5
  Pneumonia | 2.2 | 1.9
  Antibiotic use for other reasons | 8.6 | 9.3
  At least one complication and/or use of antibiotic | 16.6 | 15.4

13. Secondary Outcome: Percentage of Participants Who Required New or Increased Use of Supplemental Oxygen
Description: Percentage of participants who required new or increased use of supplemental oxygen
Time Frame: From treatment initiation to Day 28
Population: as for outcome 5
Measure: Number; unit: percentage of participants analyzed
Arm/Group | Combination Therapy | Oseltamivir Monotherapy
Number analyzed (Participants) | 314 | 312
percentage of participants analyzed | 1.91 | 1.6

14. Secondary Outcome: Percentage of Participants Who Required Hospitalization.
Description: The percentage of participants hospitalized by 28 days was estimated from the Kaplan-Meier curves.
Time Frame: From treatment initiation to Day 28
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants analyzed
Arm/Group | Combination Therapy | Oseltamivir Monotherapy
Number analyzed (Participants) | 314 | 312
percentage of participants analyzed | 4.28 [2 to 6.56] | 0.98 [-0.12 to 2.08]

15. Secondary Outcome: 28-day Mortality
Description: Number of deaths
Time Frame: From treatment initiation to Day 28
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Combination Therapy | Oseltamivir Monotherapy
Number analyzed (Participants) | 314 | 312
participants | 0 | 1

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the conduct of the study; from Day 0 to Day 28
Description: All worsening and new symptoms were evaluated as potential adverse events.If a diagnosis was clinically evident (or subsequently determined), the diagnosis, rather than the individual signs and symptoms or lab abnormalities, were recorded as the AE. All worsening laboratory values were also evaluated as potential adverse events. The DAIDS AE Grading Table (V1.0) was used.
Arm/Group | Combination Therapy | Oseltamivir Monotherapy
All-Cause Mortality (participants affected / at risk) | 0/314 | 1/312
Serious Adverse Events (participants affected / at risk) | 14/314 | 6/312
Other Adverse Events (participants affected / at risk) | 148/314 | 163/312
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Combination Therapy (N=314) | Oseltamivir Monotherapy (N=312)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Atrial tachycardia (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Delirium (Psychiatric disorders) | 0 | 1
Personality change (Psychiatric disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Combination Therapy (N=314) | Oseltamivir Monotherapy (N=312)
Diarrhoea (Gastrointestinal disorders) | 40 | 52
Nausea (Gastrointestinal disorders) | 52 | 50
Vomiting (Gastrointestinal disorders) | 34 | 22
Fatigue (General disorders) | 18 | 12
Pyrexia (General disorders) | 16 | 18
Myalgia (Musculoskeletal and connective tissue disorders) | 17 | 13
Dizziness (Nervous system disorders) | 23 | 22
Headache (Nervous system disorders) | 14 | 19
Cough (Respiratory, thoracic and mediastinal disorders) | 14 | 22
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 15 | 11
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 13 | 17
Hypertension (Vascular disorders) | 12 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No